CLINICAL TRIAL: NCT00186238
Title: High Dose Sequential Therapy and Autologous Stem Cell Rescue for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sally Arai, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT27; 73217; BMT27; NCT00186238
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Procedure: high dose chemotherapy then autologous hematopoietic cell transplant

SUMMARY:
To assess the role of autologous hematopoietic cell rescue in the treatment of multiple myeloma.

DETAILED DESCRIPTION:
To assess the toxicity and efficacy of sequentially administered high dose cyclophosphamide and VP-16 followed by total body irradiation or BCNU and high dose mephalan and autologous stem cell rescue in the treatment of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:- received cytoreduction prior to transplant

* adequate organ function Exclusion Criteria:- previous transplant
* smoldering MM or benign monoclonal gammopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1994-09; Primary Completion 2006-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Toxicity and efficacy of sequentially administered high dose chemotherapy and autologous hematopoietic cell transplantation | Patients will have a daily CBC with platelet count, and chemistries until engraftment, then as indicated clinically. Chest x-rays will be done weekly until engraftment, then as indicated clinically. Patients will be restaged for abnormal proteins (SPIE)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Arai, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States